CLINICAL TRIAL: NCT03985761
Title: Utilizing Gaming Mechanics to Optimize Telerehabilitation Adherence in Persons With Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); New Jersey Institute of Technology (Other)
Responsible Party: Principal Investigator, Gerard G Fluet DPT, PhD, Associate Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AWD00004386; 1R15HD095403-01 (NIH)
Record Dates: First submitted 2019-04-26; First posted 2019-06-14 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Stroke
Keywords: Stroke; Upper extremity; Hand; Arm; Virtual reality; Telerehabilitation; Gaming; Hemiparesis; Dexterity
MeSH Terms: conditions — Stroke; Paresis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home Telerehabilitation_Motivation Enhanced HTme (Experimental): The Home Telerehabilitation Motivation Enhanced (HTme) group will use the NJIT-HoVRS system to play a series of three games to train movement of their shoulder, elbow, wrist and fingers. The study team will set up the apparatus in their home at the initial visit and train them to use the system. After this, subjects will practice in their homes with on-line or in-person support as needed (once a week in person for the first month, and then an average of two times per month in person and two times per month on line). Subjects will be instructed to perform three of the simulations assigned to them as much as possible, but at least twenty minutes, daily for twelve weeks. The HTme group will use three simulations that will provide the user with eight to twelve levels of gradually increasing difficulty and complexity. A screen announces each level change and the graphics for each new level change substantially. Scoring opportunities increase at each new level.
  Interventions: Behavioral: Home Telerehabilitation using HoVRS
- Home Telerehabilitation_Unenhanced (HTu) (Active Comparator): The Home Telerehabilitation Motivation Enhanced (HTu) group will use the NJIT-HoVRS system to play a series of three games to train movement of their shoulder, elbow, wrist and fingers. The study team will set up the apparatus in their home at the initial visit and train them to use the system. After this, subjects will practice in their homes with on-line or in-person support as needed (once a week in person for the first month, and then an average of two times per month in person and two times per month on line). Subjects will be instructed to perform three of the simulations assigned to them as much as possible, but at least twenty minutes, daily for twelve weeks. The HTu group will use three simulations. Difficulty will be increased utilizing an adaptive control algorithm that increases difficulty based on performance. Difficulty changes are extremely incremental making them imperceptible for most subjects. Graphics and scoring do not change as difficulty level changes.
  Interventions: Behavioral: Home Telerehabilitation using HoVRS

INTERVENTIONS:
Behavioral: Home Telerehabilitation using HoVRS — The Home Virtual Rehabilitation System (HoVRS) integrates a Leap Motion controller, a passive arm support and a suite of custom designed hand rehabilitation simulations. The Leap Motion provides camera based measurement of finger joint positions, allowing for integrated virtual arm and finger training. If the patient's arm is severely impaired, a forearm orthosis that counter-balances gravity to provide graded support to the arm during activity is issued to the subject. In this study, we utilize 3 task-based simulations that train hand manipulation and arm transport. One simulation trains hand opening integrated with pronation and supination, a second trains wrist movement, by presenting targets that subjects navigate a plane over and around buildings to collect, a third simulation, trains shoulder and elbow disassociation in a horizontal plane integrated with hand opening.

SUMMARY:
This trial studies the impact of motivational strategies designed by the gaming industry on adherence to a home tele-rehabilitation program designed to improve hand function in persons with stroke. A growing literature suggests that the extended practice of challenging hand tasks can produce measurable changes in hand function in persons with stroke. Current health care delivery systems do not support this volume of directly supervised rehabilitation, making it necessary for patients to perform a substantial amount of activity at home, unsupervised. Unfortunately, adherence to unsupervised home exercise regimens is quite poor in this population. The investigator's goal is to assess the impact of several well-established game design strategies: 1) Scaffolded increases in game difficulty 2) In-game rewards 3) Quests with enhanced narrative. The investigator's will utilize these enhancements to study their impact on motivation to perform a tele-rehabilitation- based home exercise program, adherence to the program and changes in hand function. The proposed study will utilize a system of novel rehabilitation technologies designed to facilitate home exercise performance. Subjects will perform 3 simulated rehabilitation activities supported by a passive exoskeleton, an infrared camera and software that will allow subjects to exercise at home. The investigator's will investigate: 1) Differences in measures of motivation elicited by motivationally enhanced simulations and un-enhanced control versions.2) The impact of motivational enhancements on actual adherence to a tele-rehabilitation program in persons with stroke and 3) The impact of motivational enhancement on improvements in hand function achieved by these subjects. This proposal will address a critical gap in modern rehabilitation - adherence to autonomous rehabilitation programs. Patient participation in unsupervised rehabilitation is one of the assumptions underpinning our health care system. This said, no data collected to date supports that adherence is acceptable. The technology and methodology in this proposal are an important step towards leveraging extensive research and development done by the computer gaming industry into improved rehabilitation practice.

DETAILED DESCRIPTION:
1. Purpose/Specific Aims The overarching aim of this study is to provide a mechanism for patients to engage in progressive motor practice for a meaningful time period. The investigator's aim to improve on the positive outcomes demonstrated in patients in the chronic phase and the pilot work being done on patients in the acute in-patient phase post stroke to determine whether functional recovery can be further improved using a home based system.

   Aim 1: Evaluate compliance with Home-Telerehabilitation simulated hand/arm gaming activities and two computer game groups, one with motivation enhanced: Home Training Motivation Enhanced (HTme) simulations and one with non-enhanced simulations: Home Training Unenhanced (HTu) versions. Hypothesis: Participants in the HTme group will show significant compliance as compared to the control group (HTu).

   Aim 2: Evaluate the effectiveness of motivation enhanced HTme home-based virtually simulated hand/arm gaming activities for individuals with stroke as compared to a program unenhanced HTu versions of the same simulations. Hypothesis: Participants completing HTme training will exhibit significantly improved clinical, kinematic and neurophysiological outcomes as compared to the control group (HTu).

   Aim 3: Evaluate the impact of the motivation enhancements designed into computer games to provide a more enjoyable training experience. Hypothesis: Enjoyment of the games will be a more valid predictor of compliance than personal factors.
2. Background and Significance Studies have shown that sustained hand rehabilitation training is important for continuous improvement and maintenance of function following a stroke. It is unimaginably difficult to pursue education, employment and community participation without being able to independently use one's hands. The primary goal of this study is to test an exciting new technology that can be easily used in the home for long-term hand and upper extremity training. Recovery of hand function post brain injury is particularly recalcitrant to currently available interventions. To date, the best efforts of groups studying traditionally presented as well as technology-based therapeutic interventions for the hemiplegic hand and arm have produced measurable changes in motor function and motor control but fall far short of major reductions in disability.

   If the amount of therapy is critical to rehabilitation, our current institutional limitations undermine the probabilities for successful outcomes. After discharge from the inpatient stay, access to rehabilitation therapy can be difficult for some patients. This is due in part to inadequate insurance, lack of transportation, and the patient's dependence on their caregiver. Having access to long-term rehabilitation training anywhere and at any time is necessary for sub-acute and chronic patients to continuously improve their functional abilities.
3. Research Design and Methods This study will be a single blind randomized controlled trial. Subjects will be blinded to the purpose of the study. All outcome measures will be performed by a therapist blinded to group assignment. A controlled trial will be utilized to determine the additive effect of presenting rehabilitation activities in a virtual environment as compared to standard upper extremity exercise. The investigators will randomize subjects to treatment and control groups using a computerized random number generator.

   3.1. Duration of Study

   Each subject will perform a pre-study evaluation, train using one of the protocols for three months, perform a post study evaluation as well as one and six month retention evaluations.

   3.2 Study Sites Testing and initial training will take place in the Bergen Building of the Rutgers Biomedical and Health Sciences Campus in Newark. Home training will take place in subjects' homes.

   3.3 Sample Size Justification The investigators will seek sufficient power to detect a clinically significant difference in the Wolf score changes in these two pre-planned, primary comparisons. To evaluate these effects of training, we will assume a power level of .8 and a significance level of 0.05. With presumed correlation among repeated measures of 0.1 and effect size of 0.3, a sample size of 25 subjects in each of the two groups (HTme and HTu) to observe a significant effect for the first comparison (G*Power, version 3.1.5) is necessary. Although the investigators will screen for patients with homogeneous impairments, by its nature stroke is an extremely variable condition. Due to possible subject attrition, the investigators will use a total of 30 subjects in each of the two groups.

   3.4 Subject Recruitment Subjects will be recruited through flyers, stroke support groups, and clinician referrals. The investigators will assume that approximately 15-20% of the population will satisfy our inclusion criteria based on our previous experience with upper extremity rehabilitation in this population. Hence the investigators will approach 300 persons.

   3.5 Consent Procedures Example: The study will be explained to the potential subject by the study staff, the consent will be read, and their questions will be answered. If participants wish to enroll, the subject will sign the consent form. The study staff obtaining consent will also sign and date the consent form, and a copy will be given to the subject sought from each prospective subject or the subject's legally authorized representative, in accordance with federal & state law and institutional policy. If the study staff member performing the consent process identifies issues suggesting that the prospective subject may not be capable of participating in the consent process due to dementia, a Folstein Mini Mental Status will be performed. Prospective subjects screening positive for dementia will not be included in the study.

   3.5.1 Subject Costs and Compensation There are no costs for the subjects. The subjects will be paid 100$ at each of the retention tests.
4. Study Variables

   4.1 Independent Variables or Interventions

   The two computer game groups, Motivation Enhanced (HTme) and Motivation Non-Enhanced (HTu) will use the NJIT- Home Virtual Rehabilitation System (HoVRS) to play a series of computer games developed to practice movement of the hand and fingers. Subjects will first come into our lab, perform pre-tests as well as a pre-intervention training session. Then a physical therapist and engineer will set up the apparatus in subject's home and will train them on how to use the system and play the games in their home during the first week. The physical therapist and engineer will be in contact with subjects throughout the training and will visit subjects' homes as needed if problems are encountered. Additionally, the system allows the therapist to remotely monitor each day's activity.

   4.1.1 Device Description NJIT HoVRS has two sub-systems to deliver home-based training: 1) a patient based platform to provide the training and 2) a server based online data logging and reporting system. In the patient's home, a cross platform virtual reality training application runs video games (developed in the Unity 3D game engine using the language C#) on their home computer.

   4.1.11 Hardware The Leap Motion Controller (LMC) a commercially developed infrared tracking device developed for home video game control is used to capture motion of the hand and arm movement without requiring wearable sensors. The device's USB controller reads the sensor data into its own local memory and performs any necessary resolution adjustments. This data is then streamed via USB to the Leap Motion image Application Programming Interface (API). From there, we programmed the system to feed tracking data into virtual reality activities by calling the Leap Motion API.

   If the patient's arm is weak and cannot support the hand against gravity above the Leap Motion Controller, a commercially available, spring-based arm support, will be provided to the subject (Figure 1). The arm support provides 12 different levels of passive support allowing it to accommodate a wide range of patient sizes and strength levels. It requires a single setting that can be provided during the patient's initial evaluation

   4.1.1.2 Software Patients will either use their own home computer or will be provided with a computer if needed. A user-friendly Graphic User Interface (GUI) lists all of the training activities allowing patients to choose which activity they want to begin with using just one mouse click. Currently twelve games have been developed, each one designed to focus on training a specific hand or arm movement such as wrist rotation or finger individuation. All games are downloadable via HoVRS website.

   4.2 Dependent Variables: See Outcomes Measures

   4.3 Risk of Harm

   There is less than minimal risk involved. The virtual reality (VR) experiments are non-invasive and pose no obvious risk. Transient fatigue of the hand and arm are possible, but this risk is not greater than that posed by normal daily activities following a stroke.

   4.4 Potential for Benefit The benefits of taking part in this study may be: Patient may regain better use of their hand and arm. However, it is possible that patients might receive no direct personal benefit from taking part in this study.
5. Data Handling and Statistical Analysis All efforts will be made to keep subjects' personal information confidential. All subject names will be removed from the data and the data will be tagged using a coded identification (ID) number. Demographic, clinical outcome and survey data will first be recorded on paper. All kinematic and computerized performance data will be collected on computer. These computer files will be identified by the coded subject ID number. All data will be transferred to an Excel spreadsheet with subjects identified by this same ID number. Spreadsheets will be stored on a drive that is password protected. Data will only be accessible to study staff and will be retained for seven years. The link between subject identity and subject ID number will be destroyed when data collection is completed.

The primary outcome measures and all secondary outcome measures described above will be subjected to a repeated measured analysis of variance, with between-group factors Therapy Type (HTme, HTu) and within-group factor Test (Before, Post, One Month retention, Six Months Retention). Post-hoc analyses of the Therapy Type by Test interaction effects will focus on the Month 1 versus Month 6 comparison. The investigators will be quantifying training effects by comparing group means as well as by percent change in performance, and by comparing the recovery curves obtained from Tests 1-4. All clinical outcomes used are well established measures of upper extremity functional recovery with published minimum clinically important differences which will be used to evaluate the significance of our findings.

7. Reporting Results

7.1 Individual Results No disease screening data will be collected. Patient's changes on clinical tests will be shared with them during testing sessions. These sessions are conducted by licensed Physical Therapists who have training to help persons with stroke interpret clinical examination findings.

7.2 Aggregate Results Subjects will not be informed of aggregate findings.

7.3 Professional Reporting De-identified, aggregate findings will be published in professional journals and presented at scientific meetings.

ELIGIBILITY:
Inclusion Criteria:

1. unilateral stroke
2. score of 22 or greater on the Montreal Cognitive Assesment
3. Score of 1 or better on extinction and inattention portion of NIH Stroke Scale
4. Fugl-Meyer (FM) between 36-58/66 (
5. Score of 1 or better on language portion of NIHSS
6. intact cutaneous sensation (ability to detect <4.17 Newton stimulation using Semmes-Weinstein nylon filaments)

Exclusion Criteria:

Orthopedic issues that would limit the ability to perform regular upper extremity activity

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2019-09-08 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Rutgers The State University of New Jersey, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
Immediately following completion of our proposed study we will submit a de-identified data set our protocol and links to published papers based on the data set to the Centralized Open Access Rehabilitation Data Base for Stroke (SCOAR).
Supporting Information: Study Protocol
Time Frame: We will make our data available immediately after study completion. Data will remain available indefinitely.
Access Criteria: Not Applicable - Open Access
URL: http://keithlohse.github.io/SCOAR_data_viz/#

REFERENCES:
- [Background] McAuley E, Duncan T, Tammen VV. Psychometric properties of the Intrinsic Motivation Inventory in a competitive sport setting: a confirmatory factor analysis. Res Q Exerc Sport. 1989 Mar;60(1):48-58. doi: 10.1080/02701367.1989.10607413. PMID 2489825
- [Background] Hibbard JH, Stockard J, Mahoney ER, Tusler M. Development of the Patient Activation Measure (PAM): conceptualizing and measuring activation in patients and consumers. Health Serv Res. 2004 Aug;39(4 Pt 1):1005-26. doi: 10.1111/j.1475-6773.2004.00269.x. PMID 15230939
- [Background] Winstein CJ, Wolf SL, Dromerick AW, Lane CJ, Nelsen MA, Lewthwaite R, Cen SY, Azen SP; Interdisciplinary Comprehensive Arm Rehabilitation Evaluation (ICARE) Investigative Team. Effect of a Task-Oriented Rehabilitation Program on Upper Extremity Recovery Following Motor Stroke: The ICARE Randomized Clinical Trial. JAMA. 2016 Feb 9;315(6):571-81. doi: 10.1001/jama.2016.0276. PMID 26864411
- [Background] Kwakkel G. Impact of intensity of practice after stroke: issues for consideration. Disabil Rehabil. 2006 Jul 15-30;28(13-14):823-30. doi: 10.1080/09638280500534861. PMID 16777769
- [Background] Yozbatiran N, Der-Yeghiaian L, Cramer SC. A standardized approach to performing the action research arm test. Neurorehabil Neural Repair. 2008 Jan-Feb;22(1):78-90. doi: 10.1177/1545968307305353. Epub 2007 Aug 17. PMID 17704352
- [Background] Fluet GG, Patel J, Qiu Q, Yarossi M, Massood S, Adamovich SV, Tunik E, Merians AS. Motor skill changes and neurophysiologic adaptation to recovery-oriented virtual rehabilitation of hand function in a person with subacute stroke: a case study. Disabil Rehabil. 2017 Jul;39(15):1524-1531. doi: 10.1080/09638288.2016.1226421. Epub 2016 Sep 27. PMID 27669997
- [Background] Mathiowetz V, Volland G, Kashman N, Weber K. Adult norms for the Box and Block Test of manual dexterity. Am J Occup Ther. 1985 Jun;39(6):386-91. doi: 10.5014/ajot.39.6.386. PMID 3160243
- [Background] Oxford Grice K, Vogel KA, Le V, Mitchell A, Muniz S, Vollmer MA. Adult norms for a commercially available Nine Hole Peg Test for finger dexterity. Am J Occup Ther. 2003 Sep-Oct;57(5):570-3. doi: 10.5014/ajot.57.5.570. PMID 14527120
- [Background] Jurkiewicz MT, Marzolini S, Oh P. Adherence to a home-based exercise program for individuals after stroke. Top Stroke Rehabil. 2011 May-Jun;18(3):277-84. doi: 10.1310/tsr1803-277. PMID 21642065
- [Background] Miller KJ, Adair BS, Pearce AJ, Said CM, Ozanne E, Morris MM. Effectiveness and feasibility of virtual reality and gaming system use at home by older adults for enabling physical activity to improve health-related domains: a systematic review. Age Ageing. 2014 Mar;43(2):188-95. doi: 10.1093/ageing/aft194. Epub 2013 Dec 17. PMID 24351549
- [Background] Duncan PW, Wallace D, Lai SM, Johnson D, Embretson S, Laster LJ. The stroke impact scale version 2.0. Evaluation of reliability, validity, and sensitivity to change. Stroke. 1999 Oct;30(10):2131-40. doi: 10.1161/01.str.30.10.2131. PMID 10512918
- [Background] Rimmer JH, Wang E, Smith D. Barriers associated with exercise and community access for individuals with stroke. J Rehabil Res Dev. 2008;45(2):315-22. doi: 10.1682/jrrd.2007.02.0042. PMID 18566948
- [Background] Standen PJ, Threapleton K, Connell L, Richardson A, Brown DJ, Battersby S, Sutton CJ, Platts F. Patients' use of a home-based virtual reality system to provide rehabilitation of the upper limb following stroke. Phys Ther. 2015 Mar;95(3):350-9. doi: 10.2522/ptj.20130564. Epub 2014 Sep 11. PMID 25212521
- [Background] Nijenhuis SM, Prange GB, Amirabdollahian F, Sale P, Infarinato F, Nasr N, Mountain G, Hermens HJ, Stienen AH, Buurke JH, Rietman JS. Feasibility study into self-administered training at home using an arm and hand device with motivational gaming environment in chronic stroke. J Neuroeng Rehabil. 2015 Oct 9;12:89. doi: 10.1186/s12984-015-0080-y. PMID 26452749
- [Background] Wittmann F, Held JP, Lambercy O, Starkey ML, Curt A, Hover R, Gassert R, Luft AR, Gonzenbach RR. Self-directed arm therapy at home after stroke with a sensor-based virtual reality training system. J Neuroeng Rehabil. 2016 Aug 11;13(1):75. doi: 10.1186/s12984-016-0182-1. PMID 27515583
- [Background] Patel J, Qiu Q, Yarossi M, Merians A, Massood S, Tunik E, Adamovich S, Fluet G. Exploring the impact of visual and movement based priming on a motor intervention in the acute phase post-stroke in persons with severe hemiparesis of the upper extremity. Disabil Rehabil. 2017 Jul;39(15):1515-1523. doi: 10.1080/09638288.2016.1226419. Epub 2016 Sep 16. PMID 27636200
- [Background] Timmermans AA, Seelen HA, Willmann RD, Kingma H. Technology-assisted training of arm-hand skills in stroke: concepts on reacquisition of motor control and therapist guidelines for rehabilitation technology design. J Neuroeng Rehabil. 2009 Jan 20;6:1. doi: 10.1186/1743-0003-6-1. PMID 19154570
- [Background] Adamovich SV, Fluet GG, Mathai A, Qiu Q, Lewis J, Merians AS. Design of a complex virtual reality simulation to train finger motion for persons with hemiparesis: a proof of concept study. J Neuroeng Rehabil. 2009 Jul 17;6:28. doi: 10.1186/1743-0003-6-28. PMID 19615045
- [Background] Fluet GG, Merians AS, Qiu Q, Lafond I, Saleh S, Ruano V, Delmonico AR, Adamovich SV. Robots integrated with virtual reality simulations for customized motor training in a person with upper extremity hemiparesis: a case study. J Neurol Phys Ther. 2012 Jun;36(2):79-86. doi: 10.1097/NPT.0b013e3182566f3f. PMID 22592063
- [Background] Fluet GG, Merians AS, Qiu Q, Davidow A, Adamovich SV. Comparing integrated training of the hand and arm with isolated training of the same effectors in persons with stroke using haptically rendered virtual environments, a randomized clinical trial. J Neuroeng Rehabil. 2014 Aug 23;11:126. doi: 10.1186/1743-0003-11-126. PMID 25148846
- [Background] Merians AS, Fluet GG, Qiu Q, Saleh S, Lafond I, Davidow A, Adamovich SV. Robotically facilitated virtual rehabilitation of arm transport integrated with finger movement in persons with hemiparesis. J Neuroeng Rehabil. 2011 May 16;8:27. doi: 10.1186/1743-0003-8-27. PMID 21575185
- [Background] Lang CE, Macdonald JR, Reisman DS, Boyd L, Jacobson Kimberley T, Schindler-Ivens SM, Hornby TG, Ross SA, Scheets PL. Observation of amounts of movement practice provided during stroke rehabilitation. Arch Phys Med Rehabil. 2009 Oct;90(10):1692-8. doi: 10.1016/j.apmr.2009.04.005. PMID 19801058
- [Background] Lohse KR, Lang CE, Boyd LA. Is more better? Using metadata to explore dose-response relationships in stroke rehabilitation. Stroke. 2014 Jul;45(7):2053-8. doi: 10.1161/STROKEAHA.114.004695. Epub 2014 May 27. PMID 24867924
- [Background] Miller KK, Porter RE, DeBaun-Sprague E, Van Puymbroeck M, Schmid AA. Exercise after Stroke: Patient Adherence and Beliefs after Discharge from Rehabilitation. Top Stroke Rehabil. 2017 Mar;24(2):142-148. doi: 10.1080/10749357.2016.1200292. Epub 2016 Jun 23. PMID 27334684
- [Background] Simpson LA, Eng JJ, Tawashy AE. Exercise perceptions among people with stroke: Barriers and facilitators to participation. Int J Ther Rehabil. 2011 Sep 6;18(9):520-530. doi: 10.12968/ijtr.2011.18.9.520. PMID 23255881
- [Background] Rand D, Givon N, Weingarden H, Nota A, Zeilig G. Eliciting upper extremity purposeful movements using video games: a comparison with traditional therapy for stroke rehabilitation. Neurorehabil Neural Repair. 2014 Oct;28(8):733-9. doi: 10.1177/1545968314521008. Epub 2014 Feb 10. PMID 24515927
- [Background] Peters DM, McPherson AK, Fletcher B, McClenaghan BA, Fritz SL. Counting repetitions: an observational study of video game play in people with chronic poststroke hemiparesis. J Neurol Phys Ther. 2013 Sep;37(3):105-11. doi: 10.1097/NPT.0b013e31829ee9bc. PMID 23872681
- [Background] da Silva Cameirao M, Bermudez I Badia S, Duarte E, Verschure PF. Virtual reality based rehabilitation speeds up functional recovery of the upper extremities after stroke: a randomized controlled pilot study in the acute phase of stroke using the rehabilitation gaming system. Restor Neurol Neurosci. 2011;29(5):287-98. doi: 10.3233/RNN-2011-0599. PMID 21697589
- [Background] Shirzad N, Van der Loos HF. Adaptation of task difficulty in rehabilitation exercises based on the user's motor performance and physiological responses. IEEE Int Conf Rehabil Robot. 2013 Jun;2013:6650429. doi: 10.1109/ICORR.2013.6650429. PMID 24187247
- [Background] Laver KE, Lange B, George S, Deutsch JE, Saposnik G, Crotty M. Virtual reality for stroke rehabilitation. Cochrane Database Syst Rev. 2017 Nov 20;11(11):CD008349. doi: 10.1002/14651858.CD008349.pub4. PMID 29156493
- [Background] Zondervan DK, Friedman N, Chang E, Zhao X, Augsburger R, Reinkensmeyer DJ, Cramer SC. Home-based hand rehabilitation after chronic stroke: Randomized, controlled single-blind trial comparing the MusicGlove with a conventional exercise program. J Rehabil Res Dev. 2016;53(4):457-72. doi: 10.1682/JRRD.2015.04.0057. PMID 27532880
- [Background] Lum PS, Mulroy S, Amdur RL, Requejo P, Prilutsky BI, Dromerick AW. Gains in upper extremity function after stroke via recovery or compensation: Potential differential effects on amount of real-world limb use. Top Stroke Rehabil. 2009 Jul-Aug;16(4):237-53. doi: 10.1310/tsr1604-237. PMID 19740730
- [Background] Krakauer JW, Carmichael ST, Corbett D, Wittenberg GF. Getting neurorehabilitation right: what can be learned from animal models? Neurorehabil Neural Repair. 2012 Oct;26(8):923-31. doi: 10.1177/1545968312440745. Epub 2012 Mar 30. PMID 22466792
- [Background] Folstein MF, Robins LN, Helzer JE. The Mini-Mental State Examination. Arch Gen Psychiatry. 1983 Jul;40(7):812. doi: 10.1001/archpsyc.1983.01790060110016. No abstract available. PMID 6860082
- [Background] Hibbard JH, Mahoney ER, Stock R, Tusler M. Do increases in patient activation result in improved self-management behaviors? Health Serv Res. 2007 Aug;42(4):1443-63. doi: 10.1111/j.1475-6773.2006.00669.x. PMID 17610432
- [Background] Bollen JC, Dean SG, Siegert RJ, Howe TE, Goodwin VA. A systematic review of measures of self-reported adherence to unsupervised home-based rehabilitation exercise programmes, and their psychometric properties. BMJ Open. 2014 Jun 27;4(6):e005044. doi: 10.1136/bmjopen-2014-005044. PMID 24972606
- [Background] Rohafza M, Fluet GG, Qiu Q, Adamovich S. Correlation of reaching and grasping kinematics and clinical measures of upper extremity function in persons with stroke related hemiplegia. Annu Int Conf IEEE Eng Med Biol Soc. 2014;2014:3610-3. doi: 10.1109/EMBC.2014.6944404. PMID 25570772
- [Background] Merians AS, Poizner H, Boian R, Burdea G, Adamovich S. Sensorimotor training in a virtual reality environment: does it improve functional recovery poststroke? Neurorehabil Neural Repair. 2006 Jun;20(2):252-67. doi: 10.1177/1545968306286914. PMID 16679503
- [Background] Puthenveettil S, Fluet G, Qiu Q, Adamovich S. Classification of hand preshaping in persons with stroke using Linear Discriminant Analysis. Annu Int Conf IEEE Eng Med Biol Soc. 2012;2012:4563-6. doi: 10.1109/EMBC.2012.6346982. PMID 23366943
- [Derived] Fluet G, Qiu Q, Gross A, Gorin H, Patel J, Merians A, Adamovich S. The influence of scaffolding on intrinsic motivation and autonomous adherence to a game-based, sparsely supervised home rehabilitation program for people with upper extremity hemiparesis due to stroke. A randomized controlled trial. J Neuroeng Rehabil. 2024 Aug 13;21(1):143. doi: 10.1186/s12984-024-01441-7. PMID 39138516
- [Derived] Fluet G, Qiu Q, Gross A, Gorin H, Patel J, Merians A, Adamovich S. The influence of scaffolding on intrinsic motivation and autonomous adherence to a game-based, unsupervised home rehabilitation program for people with upper extremity hemiparesis due to stroke. A randomized controlled trial. Res Sq [Preprint]. 2024 Jun 7:rs.3.rs-4438077. doi: 10.21203/rs.3.rs-4438077/v1. PMID 38883760

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 48 subjects screened 15 pre-assignment screen failures due to insufficient motor or sensory function
Groups:
- Home Telerehabilitation_Motivation Enhanced HTme: 12 Weeks Training - Motivation enhanced games
- Home Telerehabilitation_Unenhanced (HTu): 12 weeks training - unenhanced, algorithm controlled games,
Period: Overall Study
Arm/Group | Home Telerehabilitation_Motivation Enhanced HTme | Home Telerehabilitation_Unenhanced (HTu)
Started | 17 | 16
Completed | 15 | 13
Not Completed | 2 | 3
Not completed — Withdrawal by Subject | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Home Telerehabilitation_Motivation Enhanced HTme | Home Telerehabilitation_Unenhanced (HTu) | Total
Number analyzed (Participants) | 15 | 13 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 11 | 21
  >=65 years | 5 | 2 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (11.1) | 55.9 (14.5) | 56.7 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 9 | 22
  Male | 2 | 4 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 13 | 11 | 24
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 13 | 10 | 23
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 13 | 28
Time since stroke in months [Mean (Standard Deviation); unit: Months] | 29 (28.8) | 63 (84) | 47.3 (64.8)
Severity of stroke as measured by Upper Extremity Fugl Meyer Assessment [Mean (Standard Deviation); unit: units on a scale] — The Upper Extremity Fugl-Meyer Assessment is a clinical scale that is a composite measure of 33 performance based items, scored 0,1 or 2. Total score reflects the sum of the 33 individual item scores. Higher scores reflect better performance.
  units on a scale | 43 (14) | 43 (12) | 43 (13)

OUTCOME MEASURES:

1. Primary Outcome: Total Intervention Time
Description: Total intervention time performed by patient during study period
Time Frame: Day one through day ninety of intervention period
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | Home Telerehabilitation_Motivation Enhanced HTme | Home Telerehabilitation_Unenhanced (HTu)
Number analyzed (Participants) | 15 | 13
Minutes | 966 [442 to 1570] | 680 [412 to 902]
Statistical Analysis 1: Comparison: Home Telerehabilitation_Motivation Enhanced HTme vs Home Telerehabilitation_Unenhanced (HTu); Test type: Superiority; p = .182, ANOVA

2. Primary Outcome: Upper Extremity Fugl Meyer Assessment
Description: Difference between post test and pretest Upper Extremity Fugl Meyer Assessment Scores. Scores between 0 and 66. The Upper Extremity Fugl-Meyer Assessment is a clinical scale that is a composite measure of 33 performance based items, scored 0,1 or 2. Total score reflects the sum of the 33 individual item scores. Higher scores reflect better performance.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Home Telerehabilitation_Motivation Enhanced HTme | Home Telerehabilitation_Unenhanced (HTu)
Number analyzed (Participants) | 15 | 13
units on a scale | 5.23 (3.2) | 6.4 (2.5)
Statistical Analysis 1: Comparison: Home Telerehabilitation_Motivation Enhanced HTme vs Home Telerehabilitation_Unenhanced (HTu); Test type: Superiority; p = .296, ANOVA

3. Primary Outcome: Intrinsic Motivation Inventory
Description: Difference between score measured three months after baseline and the score measured at baseline on the Intrinsic Motivation Inventory. Scores range = 0-84. Higher score equals higher levels of intrinsic motivation.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Home Telerehabilitation_Motivation Enhanced HTme | Home Telerehabilitation_Unenhanced (HTu)
Number analyzed (Participants) | 15 | 13
score on a scale | 5.62 (4.4) | 4.22 (5.7)
Statistical Analysis 1: Comparison: Home Telerehabilitation_Motivation Enhanced HTme vs Home Telerehabilitation_Unenhanced (HTu); Test type: Superiority; p = .483, ANOVA

4. Secondary Outcome: Average Intervention Time Per Intervention Day
Description: Average intervention time performed by the subject
Time Frame: Day one through day ninety of intervention period
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Home Telerehabilitation_Motivation Enhanced HTme | Home Telerehabilitation_Unenhanced (HTu)
Number analyzed (Participants) | 15 | 13
Minutes | 20.9 (9) | 20.9 (11)
Statistical Analysis 1: Comparison: Home Telerehabilitation_Motivation Enhanced HTme vs Home Telerehabilitation_Unenhanced (HTu); Test type: Superiority; p = .995, ANOVA

5. Secondary Outcome: Action Research Arm Test
Description: Difference between score measured three months after baseline and the score measured at baseline on the Action Research Arm Test. Range = 0 - 57. Higher scores = better function.
Time Frame: 12 weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Home Telerehabilitation_Motivation Enhanced HTme | Home Telerehabilitation_Unenhanced (HTu)
Number analyzed (Participants) | 15 | 13
score on a scale | 5.62 (4.9) | 3.47 (3.9)
Statistical Analysis 1: Comparison: Home Telerehabilitation_Motivation Enhanced HTme vs Home Telerehabilitation_Unenhanced (HTu); Test type: Superiority; p = .220, ANOVA

6. Secondary Outcome: Box and Blocks Test
Description: Difference between posttest and pretest Box and Blocks Test scores. Score reflects the number of blocks transported from one receptacle to another in sixty seconds using the stroke impaired hand. Higher scores reflect better performance.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Blocks moved in 60 seconds
Arm/Group | Home Telerehabilitation_Motivation Enhanced HTme | Home Telerehabilitation_Unenhanced (HTu)
Number analyzed (Participants) | 15 | 13
Blocks moved in 60 seconds | 3.7 (3.1) | 2.9 (3.0)
Statistical Analysis 1: Comparison: Home Telerehabilitation_Motivation Enhanced HTme vs Home Telerehabilitation_Unenhanced (HTu); Test type: Superiority; p = .538, ANOVA

7. Other Pre Specified Outcome: Stroke Impact Scale - Hand Subscale
Description: Difference between posttest and pretest score on the Stroke Impact Scales Hand Subscale. Range = 0 - 25. Higher score = better recovery. Subscales reported individually.
Time Frame: 12 weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Home Telerehabilitation_Motivation Enhanced HTme | Home Telerehabilitation_Unenhanced (HTu)
Number analyzed (Participants) | 15 | 13
score on a scale | 1.81 (2.5) | 0.82 (3.7)

8. Other Pre Specified Outcome: Stroke Impact Scale - Activities of Daily Living Subscale
Description: Difference between score measured three months after baseline and the score measured at baseline on the Stroke Impact Scales Activities of Daily Living subscale. Range = 0-50. Higher score = better recovery.
Time Frame: 12 weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Home Telerehabilitation_Motivation Enhanced HTme | Home Telerehabilitation_Unenhanced (HTu)
Number analyzed (Participants) | 15 | 13
score on a scale | 3.39 (2.2) | 1.77 (2.9)

9. Other Pre Specified Outcome: Total Training Sessions
Description: Number of training sessions performed by subject during training period
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Sessions
Arm/Group | Home Telerehabilitation_Motivation Enhanced HTme | Home Telerehabilitation_Unenhanced (HTu)
Number analyzed (Participants) | 15 | 13
Sessions | 47.7 (16.4) | 37.1 (18.4)
Statistical Analysis 1: Comparison: Home Telerehabilitation_Motivation Enhanced HTme vs Home Telerehabilitation_Unenhanced (HTu); Test type: Superiority; p = .121, ANOVA

10. Other Pre Specified Outcome: Stroke Impact Scales Participation Subscale
Description: Difference between score measured three months after baseline and the score measured at baseline on the Stroke Impact Scales Participation Subscale. Range = 0 - 40. Higher scores = higher levels of participation.
Time Frame: 12 weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Home Telerehabilitation_Motivation Enhanced HTme | Home Telerehabilitation_Unenhanced (HTu)
Number analyzed (Participants) | 15 | 13
score on a scale | 2.05 (2.5) | 1.66 (2.7)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Home Telerehabilitation_Motivation Enhanced HTme | Home Telerehabilitation_Unenhanced (HTu)
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/16
Other Adverse Events (participants affected / at risk) | 0/17 | 0/16

LIMITATIONS AND CAVEATS:
Small number of subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2024-05-13): https://cdn.clinicaltrials.gov/large-docs/61/NCT03985761/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-15): https://cdn.clinicaltrials.gov/large-docs/61/NCT03985761/SAP_001.pdf
  • Informed Consent Form (2024-05-13): https://cdn.clinicaltrials.gov/large-docs/61/NCT03985761/ICF_002.pdf